CLINICAL TRIAL: NCT02241915
Title: Microbial Sealants Do Not Decrease Surgical Site Infection for Clean Contaminated Colorectal Procedures.
Brief Title: Use of a Microbial Sealant to Reduce Surgical Site Infections.
Acronym: Integuseal
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Southern California (Other)
Responsible Party: Principal Investigator, Michael Doorly, Faculty Fellow, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HS-10-00471
Record Dates: First submitted 2014-09-13; First posted 2014-09-16 (Estimated); Last update posted 2014-09-16 (Estimated); Status verified 2014-09

CONDITIONS: Surgical Site Infection; SCIP
MeSH Terms: conditions — Surgical Wound Infection | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Microbial Sealant (Active Comparator): Integuseal (Kimberly Clark)
  Interventions: Procedure: Open Colorectal Surgery; Procedure: Laparoscopic Surgery
- Control (Sham Comparator): No microbial sealant
  Interventions: Procedure: Open Colorectal Surgery; Procedure: Laparoscopic Surgery

INTERVENTIONS:
Procedure: Open Colorectal Surgery
Procedure: Laparoscopic Surgery

SUMMARY:
Surgical site infections (SSI) are costly complications that may cause significant morbidity and increase the cost of care, particularly in colorectal surgery. Microbial sealants (MS) are a new class of wound barriers aimed at decreasing SSI, however there is only evidence of benefit in clean Class 1 procedures. Based on its success in Class 1 procedures, we hypothesized that a microbial sealant could reduce the rate of SSI by half for clean contaminated colorectal procedures (Class 2).

ELIGIBILITY:
Inclusion Criteria:

1. Nonemergent colon and/or rectal abdominal surgical procedures
2. Women of child-bearing potential must have a negative serum HCG assay prior to surgery
3. Ages ≥18 years.

Exclusion Criteria:

1. Known history of hypersensitivity to cyanoacrylate, formaldehyde or acetone products.
2. Undergoing emergency surgery (urgent surgery is allowed if informed consent is obtained and the study procedures can be performed). Emergency surgery includes cases where standard bowel preparation and other preoperative assessments cannot be done.
3. Undergoing a significant concomitant surgical procedure (e.g., Whipple & organ transplant surgery).

   The following concomitant procedures are allowed: appendectomy, cholecystectomy, oophorectomy, liver biopsy/wedge resection (but not liver resection), cystectomy.
4. History of prior laparotomy within the last 60 days of this planned procedure.
5. Planned to undergo a second laparotomy or colorectal surgical procedure (e.g. colostomy or ileostomy takedown) within 60 days of this planned first procedure.
6. Evidence preoperatively of any of the following: sepsis, severe sepsis, or septic shock (note that SIRS alone is not an exclusion criteria).6, 7
7. Preoperative severe neutropenia defined as total neutrophil count ≤500 × 106/L.
8. Current abdominal wall infection/surgical site infection from previous laparotomy/laparoscopy or for any reason.
9. Receiving antibiotic therapy within the 1 week prior to the date of surgery.
10. Preoperative evaluation suggests intra-abdominal process that might preclude full closure of the skin.
11. Preoperative serum creatinine > 3 mg/dL or renal failure requiring dialysis.
12. History of ongoing treatment (e.g. chemotherapy, radiation) for non-colorectal cancer.
13. History of major organ transplantation, including bone marrow transplantation.
14. Taking systemic steroids >10 mg prednisone daily or remicade within 2 weeks prior to surgery or a history of a current immunosuppressive condition (eg, symptomatic HIV infection), defined as a CD4 count < 200.
15. Pregnant, lactating, or of childbearing potential not practicing a birth control method with a high degree of reliability (defined in section 3.1).
16. Participation within 30 days before the start of this study in any experimental drug or device study, or currently participating in a study in which the administration of investigational drug or device within 60 days is anticipated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Incidence of SSI with and without microbial sealant. | 15 Months
  Determine the rate of SSI when microbial sealant (InteguSEAL© Kimberly-Clark) is used compared to control (no microbial sealant).

SECONDARY OUTCOMES:
Subgroup incidence of SSI with and without microbial sealant | 15 months
  Compare SSI for open vs. laparoscopy colectomy, age, BMI, diabetes and morbidity (ASA class), hospital readmission, reoperation and wound dehiscence with and without microbial sealant.

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles County/USC Medical Center, Los Angeles, California, United States